CLINICAL TRIAL: NCT01225120
Title: Amputee Gait Training Using Virtual Reality and Real-Time Feedback
Acronym: VRGAIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Jason M. Wilken PT, PhD, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2007.072t
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Abnormal Gait Kinematics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gait Training (Experimental)
  Interventions: Other: Gait Training

INTERVENTIONS:
Other: Gait Training — 12 sessions, 30 minutes of walking on treadmill with real time therapist directed feedback on gait kinematics.

SUMMARY:
The purpose of this repeated measures design gait training study is to develop and quantitatively assess the effectiveness of a virtual reality training environment using real-time feedback for modification of pelvic motion during gait.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral traumatic trans-tibial or transfemoral amputation
* Independent ambulation without an assistive device for a minimum of three months
* Ability to ambulate continuously for a minimum of 15 minutes
* Trans-femoral participants must use an ischial containment socket
* VAS Pain scores on the involved side of less than 4/10
* Sagittal plane ankle, knee and hip strength of 4 or greater on the uninvolved side as determined by manual muscle test.

Exclusion Criteria:

* Blindness
* TBI-Glascow Coma Scale score of 12 or lower at the time of injury
* Cardiac or pulmonary problems limiting physical activity
* PTSD or other psychological condition with symptoms that would be exacerbated by participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Gait Biomechanics | 3 weeks
Gait Biomechanics | immediately prior to start of 3 week training
Gait Biomechanics | Immediately post training
Gait Biomechanics | 3 weeks from initial post training

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — Director, Military Performance Lab-Center for the Intrepid
Locations (1):
- Center for the Intrepid, Fort Sam Houston, Texas, United States